CLINICAL TRIAL: NCT02111941
Title: A Pilot Study of the Safety and Immunogenicity of Folate Receptor Alpha Peptide-Loaded Dendritic Cell Vaccination in Patients With Advanced Stage Epithelial Ovarian Cancer
Brief Title: Vaccine Therapy for Patients With Stage IIIC-IV Ovarian Epithelial, Fallopian Tube, or Primary Peritoneal Cavity Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1361; NCI-2014-00713 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13-004398 (Other: Mayo Clinic Institutional Review Board); P50CA136393 (NIH)
Record Dates: First submitted 2014-04-07; First posted 2014-04-11 (Estimated); Last update posted 2025-10-31 (Actual); Status verified 2025-05

CONDITIONS: Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Tumor; Fallopian Tube Mucinous Neoplasm; Fallopian Tube Serous Neoplasm; Fallopian Tube Transitional Cell Carcinoma; Ovarian Clear Cell Cystadenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Cystadenocarcinoma; Ovarian Seromucinous Carcinoma; Ovarian Serous Cystadenocarcinoma; Ovarian Transitional Cell Carcinoma; Primary Peritoneal Serous Adenocarcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Stage IIIC Fallopian Tube Cancer; Stage IIIC Ovarian Cancer; Stage IIIC Primary Peritoneal Cancer; Stage IV Fallopian Tube Cancer; Stage IV Ovarian Cancer; Stage IV Primary Peritoneal Cancer; Undifferentiated Fallopian Tube Carcinoma; Undifferentiated Ovarian Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (vaccine therapy) (Experimental): INDUCTION PHASE: Patients receive folate receptor alpha peptide-loaded dendritic cell vaccine ID on day 1. Treatment repeats every 3 weeks for 5 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Patients receive folate receptor alpha peptide-loaded dendritic cell vaccine ID on day 1. Treatment repeats every 3 months for 7 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Multi-epitope Folate Receptor Alpha-loaded Dendritic Cell Vaccine

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Multi-epitope Folate Receptor Alpha-loaded Dendritic Cell Vaccine — Given ID
  Other Names: FRaDC Vaccine; FRalphaDC Vaccine

SUMMARY:
This pilot clinical trial studies the safety and immunogenicity of vaccine therapy in treating patients with stage IIIC-IV ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer following surgery and chemotherapy. Vaccines made from a person's peptide treated white blood cells may help the body build an effective immune response to kill tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and tolerability of folate receptor alpha dendritic cell (FRalphaDC) vaccination (folate receptor alpha-peptide loaded dendritic cell vaccine).

SECONDARY OBJECTIVES:

I. Measure time to disease recurrence of patients treated with FRalphaDCs. II. Measure overall survival of patients treated with FRalphaDCs.

TERTIARY OBJECTIVES:

I. Determine whether FRalphaDC vaccination induces an increase in the number of FRalpha-specific interleukin (IL)-17-secreting T helper (Th) cells, as determined by enzyme-linked immunosorbent spot (ELISpot).

II. Determine whether FRalphaDC vaccination induces an increase in the number of FRalpha-specific T cells that secrete interferon (IFN)gamma, tumor necrosis factor (TNF)alpha, IL-10, and granzyme B, as determined by ELISpot.

III. Determine whether FRalphaDC vaccination induces antibodies specific for FRalpha.

IV. Determine whether FRalphaDC vaccination induces a delayed type hypersensitivity (DTH) skin reaction specific for FRalpha.

V. Measure FRalpha expression in patients' primary tumors and in tumors that recur after FRalphaDC vaccine treatment (when available).

VI. Determine whether FRalphaDC vaccination is associated with changes in peripheral blood immune cell subsets.

OUTLINE: This is a dose-escalation study.

INDUCTION PHASE: Patients receive folate receptor alpha peptide-loaded dendritic cell vaccine intradermally (ID) on day 1. Treatment repeats every 3 weeks for 5 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE: Patients receive folate receptor alpha peptide-loaded dendritic cell vaccine ID on day 1. Treatment repeats every 3 months for 7 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed surgical diagnosis of stage IIIC or stage IV epithelial ovarian, fallopian tube, or primary peritoneal cancer; patients with stage III cancer must have had peritoneal metastasis beyond pelvis more than 2 cm in greatest dimension and/or regional lymph node metastasis; NOTE: Histologic confirmation of the primary tumor is required; eligible histologies include serous, endometrioid, clear cell, mucinous, transitional cell, undifferentiated, or mixed carcinoma
* Completion of cytoreductive surgery and has completed one (and only one) course of platinum-based chemotherapy (5-9 cycles) >= 4 but =< 20 weeks prior to registration; NOTE: cytoreductive surgery may have been prior to or after the first cycle of chemotherapy but must include hysterectomy and bilateral salpingo-oophorectomy, if the uterus and/or ovaries had not previously been removed; NOTE: patients may have had more than one chemotherapy regimen (ex: paclitaxel/carboplatin switched to docetaxel/carboplatin due to allergy; weekly treatment switched to every 3 week treatment due to intolerance), but may not have received a separate course of treatment for recurrent ovarian cancer (OC); NOTE: patients may receive both neoadjuvant and adjuvant chemotherapy provided both regimens are platinum-based and total 9 or fewer chemotherapy cycles
* No evidence of disease at the time of registration, including no clinical concern for disease recurrence based on each of the following:

  * No evidence of disease by history and physical exam
  * Cancer antigen (CA)125 within normal limits
  * Computed tomography (CT) abdomen/pelvis demonstrating no radiological evidence of disease performed after completion of chemotherapy =< 28 days before entering study
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L
* Platelet count >= 75 x 10^9/L
* Hemoglobin >= 8.5 g/dL
* Lymphocytes >= 0.3 x 10^9/L
* Total bilirubin =< 2 x upper limit of normal (ULN), unless patient has a documented history of Gilbert's disease, then direct bilirubin =< 1.0 mg/dL
* Aspartate transaminase (AST) =< 3 x ULN
* Creatinine =< 2.0 mg/dL
* Monocytes >= 0.25 x 10^9/L
* Able to provide informed written consent
* Expected survival > 6 months
* Willingness to return to Mayo Clinic Rochester for follow-up appointments
* Willingness to provide blood samples for immune assessment and other tests
* Willingness to undergo a tetanus vaccination

Exclusion Criteria:

* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy; NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Other uncontrolled intercurrent illness (specify)
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 3 years prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: if there is a history or prior malignancy, they must not be receiving other specific treatment for their cancer
* History of myocardial infarction =< 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Epithelial ovarian cancer of low malignant potential (borderline tumor)
* Treatment with chemotherapy, radiation therapy, or other immunotherapy =< 4 weeks prior to registration
* Immunosuppressive therapy (excluding topical steroids) for any other condition =< 4 weeks prior to registration
* Persistent fever (> 24 hours) documented by repeated measurement =< 4 weeks prior to registration
* Diagnosis of autoimmune disease, including, but not limited to:

  * Systemic lupus erythematosus (lupus)
  * Multiple sclerosis (MS)
  * Rheumatoid arthritis (RA)
  * Ankylosing spondylitis
  * Other autoimmune disease (specify)
* Use of a systemic steroid (> 5 mg prednisone daily or equivalent) =< 4 weeks prior to registration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-04-14 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLT), graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 3 weeks
  If the accrual schema is completed and there are fewer than 5 patients with a DLT, the vaccination treatment will be considered safe in this patient population.

SECONDARY OUTCOMES:
Overall survival (OS) | Number of days from study registration until death due to any cause, assessed up to 5 years
  The Kaplan-Meier method will be used to estimate the distribution of OS.
Time to disease recurrence (TDR) | Number of days from study registration until disease recurrence or death, assessed up to 5 years
  The Kaplan-Meier method will be used to estimate the distribution of TDR.

OTHER OUTCOMES:
Change in FRalpha expression | Baseline up to week 107
  Assessed using simple summary statistics (mean and 95% confidence interval.
Change in the number of FRalpha-specific IL-17-secreting Th cells | Baseline up to week 107
  Assessed using simple summary statistics (mean and 95% confidence interval.
Change in the number of FRalpha-specific T cells that secrete IFNgamma, TNFalpha, IL-10, and granzyme B | Baseline up to week 107
  Assessed using simple summary statistics (mean and 95% confidence interval.
Changes in peripheral blood immune cell subsets | Baseline up to week 107
  Assessed using simple summary statistics (mean and 95% confidence interval.
DTH skin reaction specific for FRalpha. | Up to week 104
  The percent of each category will be calculated along with a 95% confidence interval.
Induction of antibodies specific for FRalpha | Up to week 107
  The percent of each category will be calculated along with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S. Block, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials